CLINICAL TRIAL: NCT06933797
Title: Evaluation of the Changes in LRP5 and TPH1 Levels Due to Periodontal Inflammation
Brief Title: Evaluation of the Potential Effects of LRP5 and Tph1 in the Pathogenesis of Periodontal Disease Individuals With Stage III Grade B Periodontitis
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Zulal Deniz Guner, DDS, Ankara University
Other Study IDs: 36290600/03/2024; 1919B012319473 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK))
Record Dates: First submitted 2025-04-08; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Disease; Periodontitis (Stage 3); Periodontitis Stage III
Keywords: Low-density lipoprotein receptor-associated protein 5; Tryptophan Hydroxylase 1; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stage III periodontitis: Individuals exhibiting pocket depths of >3 mm in at least two non-adjacent teeth, radiographic evidence of alveolar bone loss extending to the middle or apical third of the root, and tooth loss of ≤4 due to periodontitis were classified as having Stage III periodontitis. The additional criterion for Grade B classification was defined as a % bone loss/age ratio of 0.25-1.
- Periodontally healthy: Individuals with no signs of alveolar bone loss and an overall oral bleeding score <10% were categorized as periodontally healthy.

SUMMARY:
Objectives: The aim of this study was to determine the changes in LRP5 and TPH1 levels in serum and saliva samples due to periodontal inflammation and to evaluate the relationship between these values and clinical periodontal parameters.

Methods: Saliva and serum samples were collected from 20 systemically healthy patients with Stage III periodontitis and 20 periodontally healthy control individuals. Salivary and serum LRP5 and TPH1 levels were analyzed using enzyme-linked immunosorbent assay (ELISA). Clinical periodontal parameters, including plaque index (PI), probing pocket depth (PPD), bleeding on probing (BOP), and clinical attachment level (CAL), were recorded.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,
* At least 16 permanent teeth except 3rd molars,
* Individuals who do not use orthodontic appliances,
* Individuals who are not pregnant or lactating,
* Individuals without any systemic disease that may affect periodontal health,
* Systemically healthy individuals,
* Individuals who have not used anti-inflammatory and/or anti-microbial drugs in the last 6 months,
* Individuals who have not received periodontal treatment in the last 1 year

Exclusion Criteria:

* Pregnant/lactating individuals,
* Individuals who have used anti-inflammatory and/or anti-microbial drugs in the last 6 months,
* Individuals who have undergone periodontal treatment in the last 1 year,
* Individuals with psychiatric illness,
* Individuals with any oral infection,
* Individuals with <16 teeth, excluding molars,
* Individuals with alcohol dependence,
* Individuals with active infectious disease (acute hepatitis, AIDS, tuberculosis), cancer or any systemic condition that may affect periodontal tissues,
* Individuals receiving treatment with drugs known to affect periodontal tissues (phenytoin, cyclosporine A, calcium channel blockers)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with stage III periodontitis and periodontally healthy patients admitted to Ankara University Faculty of Dentistry Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
LRP5 | 1 month
  Low-density lipoprotein (LDL) receptor-related protein 5 (LRP5) is a WNT coreceptor in the LRP superfamily involved in a wide range of biological processes including endocytosis, cellular communication, lipid homeostasis and embryonic development. The levels of LRP5 in both serum and saliva samples were determined using commercially available ELISA kits. All assays were conducted according to the manufacturers' instructions.
TPH1 | 1 month
  The inhibitory, irreversible enzyme of serotonin synthesis from intestinal cells is tryptophan hydroxylase 1 (TPH1). The levels of TPH1 in both serum and saliva samples were determined using commercially available ELISA kits. All assays were conducted according to the manufacturers' instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry,, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yadav VK, Ryu JH, Suda N, Tanaka KF, Gingrich JA, Schutz G, Glorieux FH, Chiang CY, Zajac JD, Insogna KL, Mann JJ, Hen R, Ducy P, Karsenty G. Lrp5 controls bone formation by inhibiting serotonin synthesis in the duodenum. Cell. 2008 Nov 28;135(5):825-37. doi: 10.1016/j.cell.2008.09.059. PMID 19041748
- [Background] Jiang H, Xi Y, Jiang Q, Dai W, Qin X, Zhang J, Jiang Z, Yang G, Chen Q. LRP5 Down-Regulation Exacerbates Inflammation and Alveolar Bone Loss in Periodontitis by Inhibiting PI3K/c-FOS Signalling. J Clin Periodontol. 2025 Apr;52(4):637-650. doi: 10.1111/jcpe.14112. Epub 2025 Jan 21. PMID 39837316